CLINICAL TRIAL: NCT01333579
Title: Low-frequency Transcranial Magnetic Stimulation To Enhance Motor Recovery In The Subacute Phase After Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Adriana Bastos Conforto, Professor and Neurologist, Neurostimulation Laboratory, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCT2006/55504-0
Record Dates: First submitted 2011-04-04; First posted 2011-04-12 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active rTMS (Active Comparator): 1Hz active rTMS delivered to the unaffected hemisphere
  Interventions: Other: Repetitive transcranial magnetic stimulation
- Placebo rTMS (Placebo Comparator): 1Hz placebo rTMS delivered to the vertex
  Interventions: Other: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Other: Repetitive transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation, frequency of 1Hz, once a day for ten days.

SUMMARY:
Low-frequency repetitive transcranial magnetic stimulation (rTMS) of the unaffected hemisphere (UH) transiently improves motor function in patients in the chronic phase after stroke. The goal of this study is to investigate effects on motor recovery of low-frequency rTMS of the UH, administered in the subacute phase after stroke.

DETAILED DESCRIPTION:
Stroke is a major cause of disability and worldwide. Hand motor impairment is frequent after stroke. Even mild impairments of the upper limb negatively impact disability and quality of life in these patients significantly contributes to disability. Therapeutic alternatives for hand motor rehabilitation are deeply needed.

Repetitive transcranial magnetic stimulation (rTMS) has emerged as a potential tool to improve hand motor performance after stroke. While high-frequency rTMS (HF-rTMS) often increases motor cortical excitability, LF-rTMS often has the opposite effect. Up-regulation of excitability in the affected hemisphere by HF-rTMS or down-regulation of the UH by LF-rTMS can restore the balance in inter-hemispheric inhibition and hence, facilitate movement of the paretic hand Both strategies, as well as the combination of both, have yielded encouraging results when applied in proof-of-principle, single-session studies to patients with mild hand motor impairment in the subacute and chronic stages after stroke. However, few rTMS studies included patients less than six months after stroke, and effects of LF-rTMS of the unaffected hemisphere in patients with severe motor impairment in the subacute phase have not been yet reported.

The investigators opted for a novel approach to enhance hand motor recovery, by examining feasibility, safety and preliminary efficacy of either active or sham LF-rTMS of the UH or sham rTMS as add-on therapies to outpatient customary rehabilitation, to patients with mild to severe hand paresis, within 5-45 days after unilateral ischemic stroke. The investigators hypothesize that, at this stage, LF-rTMS will be feasible even in patients with severe motor deficits, will have minimal adverse events and will enhance effects of customary rehabilitation on hand motor performance.

ELIGIBILITY:
Inclusion Criteria:

* First-ever ischemic stroke in the internal carotid artery territory confirmed by CT or MRI, 5-45 days before, leading to contralateral hand weakness
* Age, 18-80 years

Exclusion Criteria:

* Cardiac pacemaker
* Pregnancy
* Implantable medication pump
* Intracranial hypertension
* History of seizures
* Metal in the head
* Decompressive surgery
* Other neurological diseases
* Shoulder pain
* Joint deformity in the paretic upper limb
* Severe chronic disease such as end-stage cancer or end-stage renal failure
* Inability to provide informed consent due to severe language or cognitive impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-02; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Motor function of the paretic hand evaluated with the Jebsen-Taylor test | Baseline, two weeks, 1 month, 3 and six months after end of treatment
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Baseline, two weeks, 1 month, 3 and six months after end of treatment
Number of patients able to comply with the protocol | Baseline, two weeks, 1 month, 3 and six months after end of treatment

SECONDARY OUTCOMES:
Force of the paretic hand | Baseline, two weeks, 1 month, 3 and six months after end of treatment
Fugl-Meyer evaluation of motor performance (upper limb) | Baseline, two weeks, 1 month, 3 and six months after end of treatment
Disability evaluated with the modified Rankin scale | Baseline, two weeks, 1 month, 3 and six months after end of treatment
Functional Independence Measure | Baseline, two weeks, 1 month, 3 and six months after end of treatment
Neurological impairment evaluated with the NIH Stroke Scale | Baseline, two weeks, 1 month, 3 and six months after end of treatment
Measures of corticomotor excitability evaluated with transcranial magnetic stimulation | Baseline, two weeks, 1 month, 3 and six months after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Conforto, MD, PhD, Principal Investigator — HC/FMUSP/Fundação Faculdade de Medicina
Locations (1):
- Laboratório de Neuroestimulação, HC/FMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Anjos SM, Cohen LG, Sterr A, de Andrade KN, Conforto AB. Translational neurorehabilitation research in the third world: what barriers to trial participation can teach us. Stroke. 2014 May;45(5):1495-7. doi: 10.1161/STROKEAHA.113.003572. Epub 2014 Mar 18. PMID 24643406